CLINICAL TRIAL: NCT04940000
Title: Evaluation of the Interest of a Video-assisted Remote Speech Therapy Consultation in Patients With ORL Cancer (TELE ORTHOPHONIE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21VADS03
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: ORL Cancer
Keywords: Video-Assisted Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient with T3-T4 ORL cancer, relevant to surgery and/or radiotherapy and/or chemotherapy. (Experimental)
  Interventions: Other: Patient managed at the IUCT-O and by a private speech therapist (near the patient's home).

INTERVENTIONS:
Other: Patient managed at the IUCT-O and by a private speech therapist (near the patient's home). — Each patient included will have a video-assisted remote speech therapy consultation with a private speech therapist (near the patient's home) and the expert speech therapist of IUCT-O center.
  At the end of this video consultation, the patient and the private speech therapist will be asked to complete a satisfaction questionnaire.

SUMMARY:
Interventional, prospective, single-centre study aimed to evaluate the impact of a video-assisted remote speech therapy consultation in relation to the complexity and specificity of the care of patients with ORL cancer. Three indications will be studied: phonation problems, swallowing problems and other problems.

The study will be conducted on a population of patients with T3, T4 ORL cancer requiring speech therapy.

Each patient included will have a video-assisted speech therapy consultation with a private speech therapist and an expert speech therapist. At the end of this video consultation, the patient and the private speech therapist will be asked to complete a satisfaction questionnaire.

At the follow-up visit following the video-assisted consultation, the patient will have completed participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at study entry.
2. Patient with carcinological pathology of the VADS, relevant to surgery and/or radiotherapy and/or chemotherapy.
3. Patient managed at the IUCT-O and by a private speech therapist (near the patient's home).
4. Patient affiliated to a Social Security system in France.
5. Patient having signed informed consent prior to inclusion in the study and prior to any specific study procedure.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Any psychological, familial, geographical or sociological condition that does not allow for compliance with the medical follow-up and/or procedures foreseen in the study protocol.
3. Patients deprived of their liberty or under legal protection (guardianship and tutorship, safeguard of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
The rate of patients for whom tele-therapy will be considered successful. | 12 months for each patient

SECONDARY OUTCOMES:
The rate of patients with full or partial resolution of speech-language pathology at the end of the telecare consultation. | 12 months for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, France